CLINICAL TRIAL: NCT05637814
Title: Dynamic Critical Congenital Heart Screening With Addition of Perfusion Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1933258
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease
Keywords: Machine Learning Algorithm; Pulse Oximetry
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Non-invasive measurements of oxygenation and perfusion will be measured with pulse oximeters and a machine learning algorithm to improve sensitivity of CCHD screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpO2 and PIx Measurement (Experimental): Non-invasive measurements of oxygenation (SpO2) and perfusion (PIx) will be measured with pulse oximeters and a ML CCHD screening algorithm will be assigning a prediction every minute.
  Interventions: Diagnostic Test: SpO2/PIx Measurement and ML Algorithm

INTERVENTIONS:
Diagnostic Test: SpO2/PIx Measurement and ML Algorithm — Right upper and any lower extremity oxygen saturation (SpO2) and perfusion index (PIx) will be measured and an online ML inference model will be used to classify a newborn as healthy versus CCHD as new pulse oximetry data is collected.

SUMMARY:
The purpose of this study is to implement and externally validate an inpatient ML algorithm that combines pulse oximetry features for critical congenital heart disease (CCHD) screening.

DETAILED DESCRIPTION:
The study will externally validate an algorithm that combines non-invasive oxygenation and perfusion measurements as a screening tool for CCHD. In a previous study, the investigators created an algorithm that combines non-invasive measurements of oxygenation and perfusion over at least two measurements using machine learning (ML) techniques. The prior model was created and tested using internal validation (k-fold validation). Thus, the investigators will test the model on an external sample of patients to test generalizability of the model. Additionally, the team will trial a repeated measurement for any "failure" of the screen to assess impact on the false positive rate. Study team will also use repeated pulse oximetry measurements (up to 4 total and including measurements after 48 hours of age, which may be done outpatient) to create a new algorithm that incorporates new data over time. The central hypothesis is that the addition of non-invasive perfusion measurements will be superior to SpO2-alone screening for CCHD detection and a model that incorporates repeated measurements will enhance detection of CCHD while preserving the specificity.

ELIGIBILITY:
Inclusion Criteria:

* Age < 22 days
* Fetuses suspected to have congenital heart disease
* Newborns with suspected/confirmed critical congenital heart disease
* Asymptomatic newborn undergoing SpO2 screening for CCHD

Exclusion Criteria:

* Echocardiogram completed prior to enrollment as the newborn would then no longer be considered "asymptomatic undergoing SpO2 screening for CCHD"
* For Newborns with confirmed/suspected congenital heart disease (CHD): a) Patent ductus arteriosus and/or atrial septal defect/patent foramen ovale without other defects, b) Corrective cardiac surgical or catheter intervention performed before enrollment or c) Current infusions of vasoactive medications other than prostaglandin therapy.

Ages: 0 Minutes to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve for receiver operating characteristics for critical congenital heart disease using ML inpatient algorithm. | Through study completion, an average of 4 years
  Receiver operating characteristics reflect a combination of sensitivity and specificity of a test. The investigators will identify the true positive and true negative rates for CCHD by confirming health status to a minimum of 2 months of age. The investigators will also utilize birth defect and death registries for missing infants.

SECONDARY OUTCOMES:
Sensitivity for critical congenital heart disease using ML inpatient algorithm (0-24 hours and 24-48 hours) | Through study completion, an average of 4 years
  The investigators will identify the true positive rate for CCHD by confirming health status to a minimum of 2 months of age. CCHD will be defined based on echocardiogram or parent report if echocardiogram not present. The investigators will also utilize birth defect and death registries for missing infants.
Specificity for critical congenital heart disease using ML inpatient algorithm (0-24 hours and 24-48 hours) | Through study completion, an average of 4 years
  The investigators will identify the true negative rate by confirming health status to a minimum of 2 months of age. CCHD will be defined based on echocardiogram or parent report if echocardiogram not present. The investigators will also utilize birth defect and death registries for missing infants.
Area under the curve for receiver operating characteristics for critical congenital heart disease using dynamic ML algorithm | Through study completion, an average of 4 years
  Receiver operating characteristics reflect a combination of sensitivity and specificity of a test. The investigators will identify the true positive and true negative rates for CCHD by confirming health status to a minimum of 2 months of age. The investigators will also utilize birth defect and death registries for missing infants.
Sensitivity for critical congenital heart disease using dynamic ML algorithm | Through study completion, an average of 4 years
  The investigators will identify the true positive rate for CCHD by confirming health status to a minimum of 2 months of age. CCHD will be defined based on echocardiogram or parent report if echocardiogram not present. The investigators will also utilize birth defect and death registries for missing infants.
Specificity for critical congenital heart disease using dynamic ML model | Through study completion, an average of 4 years
  The investigators will identify the true negative rate by confirming health status to a minimum of 2 months of age. CCHD will be defined based on echocardiogram or parent report if echocardiogram not present. The investigators will also utilize birth defect and death registries for missing infants.
Sensitivity for critical coarctation of the aorta using dynamic ML algorithm | Through study completion, an average of 4 years
  Critical coarctation of the aorta is the most commonly missed CCHD. The investigators will identify the true positive rate by confirming health status to a minimum of 2 months of age. The investigators will also utilize birth defect and death registries for missing infants.

OTHER OUTCOMES:
Frequency of repeated inpatient ML measurements | Through study completion, an average of 4 years
  If a newborn has an initial "fail" during the inpatient ML screening algorithm, then 1 repeated measurement will occur within 3 hours after waiting at least 30 minutes. If the next repeated measurement is a "fail" then the final classification assigned will be a "fail." If the repeat measurement is a "pass" the final classification will be a "pass." To gauge impact on nursing time for repeated measurements, The investigators will quantify how often these repeated measurements occur.
Feasibility: Number of minutes needed to obtain simultaneous artifact free hand and foot measurements such that all pulse oximetry features can be included. | Through study completion, an average of 4 years
  In order to incorporate the radiofemoral delay component of the pulse oximetry features, the hand and foot waveforms need to be artifact free simultaneously. The pulse oximetry device will give a result every minute to give the investigators an idea on how long it may take to reach simultaneously artifact free waveforms.
Feasibility: Number of outpatient pulse oximetry measurements obtained | Through study completion, an average of 4 years
  Pulse oximetry measurements are not currently conducted in the outpatient setting. Thus, the investigators will assess feasibility for future trials based on how many outpatient measurements are obtained versus missed in the study protocol.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis Medical Center, Davis, California
  - Cohen Children's Medical Center, Queens, New York
  - University of Utah Health Care, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No